CLINICAL TRIAL: NCT06758960
Title: Biological Evolution of HELLP Syndrome
Brief Title: Analysis of Biological Progression and Regression of HELLP Syndrome in Time
Status: Recruiting | Type: Observational
Sponsor: CHU Mohammed VI Marrakech (Other)
Responsible Party: Principal Investigator, Meryem Essafti, Assistant Professor, CHU Mohammed VI Marrakech
Other Study IDs: 67/2024
Record Dates: First submitted 2024-12-15; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: HELLP Syndrome; Preeclampsia
Keywords: Preeclampsia; HELLP syndrome; Thrombocytopenia; Maternal mortality
MeSH Terms: conditions — HELLP Syndrome; Pre-Eclampsia; Thrombocytopenia; Maternal Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Prospective observational study about progression and regression of biological parameters of HELLP syndrome

DETAILED DESCRIPTION:
Data collection included a comprehensive review of pathological histories, identification of complications based on clinical presentation, daily monitoring of biological parameters, documentation of transfusion events, recording of corticosteroid administration according to gestational age, and detailed reporting of extraction and analgesia techniques.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are admitted to the maternal ICU for a biological HELLP syndrome

Exclusion Criteria:

* Patients whose biological presentation was attributable to other conditions, such as microangiopathies or leukemia.
* Patients who benefited from plasma exchange therapy

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — FEMALE
Study Population: Pregnant patients admitted to the maternal ICU from the Obstetrics Emergency department of marrakesh
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Platelets count | Up to 10 days
  Platelets count will be monitored daily before and after delivery

SECONDARY OUTCOMES:
Concentration of Lactate dehydrogenase | Up to 10 days
  Monitored daily before and after delivery
Concentration of Liver enzymes | Up to 10 days
  daily monitoring of alkaline phosphatase, alanine transaminase before and after delivery

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Essafti, Assistant Professor, Study Director — CHU Mohammed VI Marrakech
Locations (1):
- CHU Mohammed VI of Marrakech, Marrakesh, Marrakech - Safi, Morocco

IPD SHARING:
Plan to Share IPD: Yes
All data collected throughout the trial will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 3 months and ending 1 year after the publication of results

REFERENCES:
- [Background] Martin JN Jr, Blake PG, Lowry SL, Perry KG Jr, Files JC, Morrison JC. Pregnancy complicated by preeclampsia-eclampsia with the syndrome of hemolysis, elevated liver enzymes, and low platelet count: how rapid is postpartum recovery? Obstet Gynecol. 1990 Nov;76(5 Pt 1):737-41. doi: 10.1097/00006250-199011000-00001. PMID 2216215
- [Background] Martin JN Jr, Blake PG, Perry KG Jr, McCaul JF, Hess LW, Martin RW. The natural history of HELLP syndrome: patterns of disease progression and regression. Am J Obstet Gynecol. 1991 Jun;164(6 Pt 1):1500-9; discussion 1509-13. doi: 10.1016/0002-9378(91)91429-z. PMID 2048596

DOCUMENTS (2):
  • Study Protocol (2024-12-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT06758960/Prot_000.pdf
  • Informed Consent Form (2024-12-14): https://cdn.clinicaltrials.gov/large-docs/60/NCT06758960/ICF_001.pdf